CLINICAL TRIAL: NCT04250389
Title: Microcirculatory Effects of Methylene Blue in Vasoplegic Shock After Cardiopulmonary Bypass: a Pilot Study
Brief Title: Microcirculatory Effects of Methylene Blue
Acronym: MAGIC BLUE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_MAGICBLUE
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Acute Circulatory Failure
Keywords: Methylene Blue
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with VS receiving methylene blue infusion: The studied population will be all patients receiving methylene blue for refractory vasoplegic shock (VS) after Cardiopulmonary Bypass (CPB). Refractory VS is defined as follow: a dose of norepinephrine > 0.5µg/kg/min to obtain a mean arterial pressure of 65-75 mmHg with a normal or increase cardiac (> 2 L.min-1.m-2). Patients will be included in the investigator's 20-bed adult cardiothoracic intensive care unit (ICU) in a tertiary teaching hospital (Hopital Cardiologique Louis Pradel, Hospices Civils de Lyon).
  Interventions: Other: Hemodynamic assessment (micro and macrocirculatory)

INTERVENTIONS:
Other: Hemodynamic assessment (micro and macrocirculatory) — Each of the variable related to macro- and microcirculatory will be evaluated before and one hour after start of MB infusion.
  Macrocirculatory parameters will include :
  * Mean, systolic, diastolic arterial, heart rate (HR)
  * Cardiac output (CO), sequential vascular response (SVR) and stroke volume (obtained with transthoracic echocardiography or transpulmonary thermodilution catheter if available).
  * A passive leg raising (PLR) test will be performed before and one hour after MB infusion. Patients will be classified as fluid responder if they had a CO of at least 10% after PLR.
  Microcirculatory parameters will include :
  * Cutaneous and gingival refill time
  * Tissue oxygen saturation combined with vascular occlusion test (VOT)
  * Video microscopy measurements of the sublingual microcirculation
  * Metabolic variables: Arterial blood gases including arterial lactate and central venous blood gases.

SUMMARY:
International guidelines recommend Methylene Blue (MB) as a second-line drug in the treatment of norepinephrine refractory vasoplegic shock (VS) after Cardiopulmonary Bypass CPB. Macrocirculatory effects of MB in this setting are now well established but microcirculatory effects of MB remain unknown.

The purpose of this study is to assess the micro vascular effects of a single administration of methylene blue (1.5 mg/kg over 30 minutes) for norepinephrine-refractory VS post CPB.

Microcirculatory effect will be monitored before and one hour after MB infusion through cutaneous refill time, video microscopy measurements of the sublingual microcirculation and tissue oxygen saturation combined with vascular occlusion test (VOT).

ELIGIBILITY:
Inclusion Criteria:

* patients receiving methylene blue prescribed by the clinician in charge of the patient
* patient receiving a dose of norepinephrine > 0.5µg/kg/min
* normal or increase cardiac (> 2 L.min-1.m-2) at the time of inclusion
* vasoplegic syndrome post cardiopulmonary bypass for cardiac surgery

Exclusion Criteria:

* the need for hemodynamic intervention during the time of study (fluid resuscitation, introduction of inotropic or vasopressor support, change in inotropic support dose)
* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving methylene blue for refractory vasoplegic shock (VS) in intensive care unit after Cardiopulmonary Bypass CPB. Refractory VS was defined as follow: a dose of norepinephrine > 0.5µg/kg/min to obtain a mean arterial pressure of 65-75 mmHg with a normal or increase cardiac (> 2 L.min-1.m-2).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in tissue oxygenation (resaturation speed expressed as %/sec) during the vessel obstruction test. | one hour after the start of methylene blue infusion
  The resaturation speed during reperfusion is defined as maximum StO2 - minimum StO2 /time of reperfusion. Tissue oxygen saturation (StO2) will be measured by near-infrared reflectance spectroscopy (NIRS) optode applied to the medial surface of the left or right forearm, 5 cm below the elbow. The sensor will be connected to the four-wavelength O3 Regional Oximetry device (Masimo Incorporation). All StO2 values will be recorded continuously and read every second. Data will be recorded online, transferred to a laptop with a specific software designed by Masimo (Masimo Instrument Configuration Tool (MICT) Version 1.0.4.9), and stored for further analysis. After completion of a baseline set of measurements for each patient, a vascular occlusion test (VOT) will be then perform using a manual pneumatic cuff inflator (Spengler SAS, Antony, France) positioned at the upper extremity of the ipsilateral upper limb.

SECONDARY OUTCOMES:
Video microscopy measurements of the sublingual microcirculation | one hour after the start of methylene blue infusion
  Proportion of Perfused Vessel (PPV), Total Vessel Density (TVD), Perfused Vessel Density (PVD), Microcirculatory Flow Index (MFI) and heterogeneity index will be reported. Video microscopy measurements will be collected before and one hour after the beginning of MB infusion.
Cutaneous and gingival refill time | one hour after the start of methylene blue infusion
  Five consecutive cutaneous recoloration time (CRT) acquisitions on the thorax and five consecutive gingival recoloration time (GRT) acquisitions will be made after calibrated compression of the skin and the gingiva. These measurements will be collected before and one hour after the beginning of MB infusion.
Metabolic variables | one hour after the start of methylene blue infusion
  Arterial blood gases including arterial lactate and central venous blood gases will be withdrawn before and one hour after the beginning of MB infusion concomitantly to measurement of cardiac output to allow calculation of oxygen delivery (DO2), oxygen uptake (VO2), oxygen extraction ratio (ER), venous-to-arterial difference in carbon dioxide partial pressure (PCO2gap), modified respiratory quotient (RQ modified) and ratio of central venous-to-arterial carbon dioxide content to arteriovenous oxygen content (DavCO2/DavO2).

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'anesthesie reanimation, Hôpital cardiologique Louis Pradel, Bron, France

REFERENCES:
- [Derived] Maurin C, Portran P, Schweizer R, Allaouchiche B, Junot S, Jacquet-Lagreze M, Fellahi JL. Effects of methylene blue on microcirculatory alterations following cardiac surgery: A prospective cohort study. Eur J Anaesthesiol. 2022 Apr 1;39(4):333-341. doi: 10.1097/EJA.0000000000001611. PMID 34610607